CLINICAL TRIAL: NCT02924584
Title: THE TREATMENT FOR RECURRENT FEMALE BREAST CANCER AFTER INITIAL ENDOCRINE THERAPY AMONG TAIWANESE POPULATION
Brief Title: Clinical Outcome Of Hormonal Receptor Positive, Her-2 Negative Breast Cancer In Taiwan
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481066; NCT02924584 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: ER/PR(+), Her2(-) Breast Cancer
Keywords: hormonal receptor positive, human epidermal growth factor receptor 2 negative, breast cancer, aromatse inhibitor, overall survival, prevalence
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Breast cancer is the most common cancer in Taiwanese women. Most of them were diagnosed in relatively early stages. Only 700 metastatic breast cancer were registered in Official Cancer Registration 2012, while more than11,305 were registered as early breast cancer. With broadly application of aromatase inhibitors, hormonal-receptor-positive breast cancer patients can survive longer and longer. However, there is no prevalence of metastatic breast cancer can be available yet. NHIA database coverage is more than 90% population in Taiwan, thus it can be an appropriate surrogate of prevalence. In this retrospective database analysis, we will explore the real world experience on aromatase inhibitor use for breast cancer in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* hormonal receptor positive, human epidermal growth factor receptor 2 negative breast cancer

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: hormonal receptor positive, human epidermal growth factor receptor 2 negative breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
clinical use of aromatase inhibitors in breast cancer | base line, up to 60 months
  duration of treatment

SECONDARY OUTCOMES:
prevalence | base line up to 60 months
  The prevalence of metastatic breast cancer with positive hormonal receptors with routine practice in Taiwan.
dose exposure | base line, up to 60 months
  The dosage pattern of breast cancer with positive hormonal receptors with routine practice in Taiwan.
overall survival | base line, up to 60 months
  The overall survival of metastatic breast cancer with positive hormonal receptors with routine practice in Taiwan.
treatment cost | base line, up to 60 months
  The treatment cost of metastatic breast cancer with positive hormonal receptors with routine practice in Taiwan.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481066